CLINICAL TRIAL: NCT00000980
Title: Single-Blind Efficacy Evaluation of Intravenous Spiramycin in Subjects With AIDS-Related Cryptosporidial Diarrhea
Brief Title: A Study of Spiramycin in the Treatment of Patients With AIDS-Related Diarrhea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhone-Poulenc Rorer (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 113; FDA 28A; CCB-301
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-10

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: Single-Blind Method; Spiramycin; AIDS-Related Opportunistic Infections; Injections, Intravenous; Cryptosporidiosis; Diarrhea; Drug Evaluation; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; AIDS-Related Opportunistic Infections; Diarrhea; Acquired Immunodeficiency Syndrome | interventions — Spiramycin

INTERVENTIONS:
Drug: Spiramycin

SUMMARY:
To determine the safety and effectiveness of intravenous spiramycin in patients with AIDS-related cryptosporidial diarrhea.

Spiramycin, a macrolide antibiotic, has been studied in the United States for the treatment of cryptosporidial diarrhea. Some reports suggest that spiramycin is useful in improving the symptoms of cryptosporidial diarrhea in some patients. Results of one study, however, showed no significant difference between spiramycin and placebo (inactive medication). A later study indicated that the absorption of spiramycin is significantly decreased when food is present. Thus, the results of the trial may have been due to poor absorption of spiramycin.

DETAILED DESCRIPTION:
Spiramycin, a macrolide antibiotic, has been studied in the United States for the treatment of cryptosporidial diarrhea. Some reports suggest that spiramycin is useful in improving the symptoms of cryptosporidial diarrhea in some patients. Results of one study, however, showed no significant difference between spiramycin and placebo (inactive medication). A later study indicated that the absorption of spiramycin is significantly decreased when food is present. Thus, the results of the trial may have been due to poor absorption of spiramycin.

Patients are observed for 3 days to establish baseline conditions. They are informed that the treatment period is 21 days during which they receive 15 days of spiramycin and 6 consecutive days of placebo; they are not told which 6-day period they receive placebo. All patients receive 15 days of spiramycin. Patients who do not have a favorable response are treated with a higher dose of spiramycin for an additional 15 days. Responders at either dose are followed weekly for 4 weeks. Should a relapse occur, patients receive an additional 15 days of therapy, at the dose of spiramycin that initially produced a response, following reestablishment of a baseline with 6 days of placebo. Nonresponders to the higher dose are taken off the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Vitamin supplements.
* Zidovudine (AZT) for patients previously taking AZT. However, dosing with spiramycin should be delayed until the dose of AZT has stabilized. The dose may be decreased for AZT-associated toxicity.

Allowed for diarrhea:

* Loperamide hydrochloride capsules (2 mg) or loperamide hydrochloride liquid (1 mg/5 ml).

Allowed for nausea:

* Sucralfate and metoclopramide hydrochloride.

Allowed for vomiting:

* Prochlorperazine and trimethobenzamide hydrochloride.
* Allowed as prophylaxis for Pneumocystis carinii pneumonia (PCP):
* Aerosolized pentamidine.

Patients must have:

* A diagnosis of AIDS according to the CDC.
* Chronic diarrhea.
* Presence of Cryptosporidium oocysts in stool specimen. Patients or a legally authorized representative must sign an informed consent form. Diet will be lactose free, maximum 7 g fat/day with unlimited calorie intake. Patients who require total parenteral nutrition will also be allowed oral intake.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Grade 4 (for hematologic) or Grade 3 (for all other) toxicity.
* Known sensitivity to macrolide antibiotics.
* Presence of other diarrhea-causing pathogens.
* Active opportunistic infection requiring systemic antimicrobial therapy.
* Toxicity grades according to NIAID toxicity scale for adults.

Concurrent Medication:

Excluded:

* Other investigational drugs.
* Cancer chemotherapy.
* Alpha interferon.
* Other immunomodulating agents.
* Other macrolide antibiotics.
* Trimethoprim / sulfamethoxazole.
* Ganciclovir.
* H2 blockers and AL-721.
* Medications known to cause gastrointestinal irritation or alteration of gastrointestinal motility or absorption should be avoided if possible.
* Zidovudine (AZT) therapy may not be initiated and the dose may not be increased during the study.

Patients with the following are excluded:

* Grade 4 (for hematologic) or Grade 3 (for all other) toxicity.
* Known sensitivity to macrolide antibiotics.
* Presence of other diarrhea-causing pathogens.
* Active opportunistic infection requiring systemic antimicrobial therapy.
* Toxicity grades according to NIAID toxicity scale for adults.

Prior Medication:

Excluded within 7 days of study entry:

* Investigational drugs.

Excluded within 14 days of study entry:

* Cancer chemotherapy.
* Alpha interferon.
* Other immunomodulating agents.
* Other macrolide antibiotics.
* Trimethoprim / sulfamethoxazole.
* Ganciclovir.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25

CONTACTS AND LOCATIONS:
Overall Officials: R Soave, Study Chair
Locations (7):
- United States (7):
  - Kaiser Permanente Med Ctr, San Diego, California
  - Johns Hopkins Univ School of Medicine, Baltimore, Maryland
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Nelson Tebedo Community Clinic, Dallas, Texas